CLINICAL TRIAL: NCT07234006
Title: EFFECT OF NEUROFEEDBACK-MINDFULNESS TECHNIQUES ON ANXIETY, STRESS, AND ACADEMIC PERFORMANCE OF NURSING STUDENTS
Brief Title: Neurofeedback-mindfulness Techniques on Anxiety, Stress, and Academic Performance of Nursing Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, José Ignacio Recio Rodriguez, Doctor, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IBYP25/034
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Anxiety; Stress; Academic Performance
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No intervention (Other): No intervention
  Interventions: Other: No intervention
- NEUROFEEDBACK-MINDFULNESS (Experimental): Neurofeedback-Assisted Mindfulness Training Program
  Interventions: Behavioral: NEUROFEEDBACK-MINDFULNESS

INTERVENTIONS:
Behavioral: NEUROFEEDBACK-MINDFULNESS — The Neurofeedback-Assisted Mindfulness Training sessions will be given to the intervention group participants after randomization. Each session will vary in length depending on the session, but will last a maximum of 20 minutes.
  A total of 20 sessions will be held at the participant's home, preferably in the afternoon, at a rate of 5 sessions per week for 4 weeks after randomization. The organization of the sessions is described in the following table of this study's protocol.
  Arms: NEUROFEEDBACK-MINDFULNESS
Other: No intervention — No intervention
  Arms: No intervention

SUMMARY:
In today's society, anxiety and stress are prevalent emotional responses in mental health globally, significantly affecting students' well-being and academic performance. In particular, undergraduate nursing students face high levels of these problems due to the heavy academic workload and demands of their training, especially during exam periods. The need for concentration, emotional management, and decision-making under pressure contribute to the prevalence of these disorders, impacting both their quality of life and academic performance.

Despite the existence of multiple strategies and techniques for managing these issues, it is still necessary to continue exploring innovative alternatives that complement traditional interventions. For this reason, this project aims to evaluate the effectiveness of mindfulness-neurofeedback as a treatment to reduce stress and anxiety in nursing students, with the goal of providing scientific evidence on this intervention. This brain training technique is presented as a promising option, based on the modulation of brain activity, with the potential to improve emotional regulation and concentration in the educational setting.

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled in the nursing degree at the University of Salamanca
* Aged between 18 and 45 years
* Willing to voluntarily participate in the study and sign the informed consent form.

Exclusion Criteria:

* History of serious psychiatric disorders in the 6 months prior to inclusion in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-11-21 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Mean of the Depression, anxiety and stress scale at 4 weeks | From enrollment to the end of treatment at 4 weeks
  Zero is equivalent to no symptoms and 63 indicates the worst possible symptoms
Change from Baseline in the Mean Academic performance score at 4 weeks | From enrollment to the end of treatment at 4 weeks
  Zero is equivalent to the best academic performance and 40 indicates the worst academic performance

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No